CLINICAL TRIAL: NCT06217003
Title: A Phase II Clinical Study of Trilaciclib Combined With Chemotherapy for Perioperative Treatment of Osteosarcoma
Brief Title: Trilaciclib Combined With Chemotherapy for Perioperative Treatment of Osteosarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSKY028
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Osteosarcoma
Keywords: Osteosarcoma; Perioperative period; Trilaciclib; Chemotherapy
MeSH Terms: conditions — Osteosarcoma | interventions — trilaciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- trilaciclib (Experimental): Screening of eligible subjects for inclusion and application of trilaciclib before undergoing perioperative chemotherapy
  Interventions: Drug: Trilaciclib

INTERVENTIONS:
Drug: Trilaciclib — Preoperative application of trilaciclib during perioperative chemotherapy

SUMMARY:
This study is a prospective, single arm phase II study aimed at evaluating the efficacy and safety of trilaciclib before perioperative chemotherapy in patients with osteosarcoma.

DETAILED DESCRIPTION:
This study is a prospective, single arm phase II study aimed at evaluating the efficacy and safety of Trilaciclib before perioperative chemotherapy in patients with osteosarcoma.Patients diagnosed by pathology and evaluated by surgeons as having non metastatic resectable osteosarcoma, after signing informed consent, will be screened for eligible subjects to receive a treatment regimen of tralazilide before perioperative chemotherapy;

The study will include 20 participants who will receive the following design scheme:

During the preoperative neoadjuvant therapy period, the subjects will receive two cycles of preoperative neoadjuvant therapy:Trilaciclib is administered daily within 4 hours before chemotherapy, 240mg/m2, intravenously; The chemotherapy regimen is MAP regimen (doxorubicin 75mg/m2, cisplatin 120mg/m2, methotrexate 8-12g/m2); Recombinant human endostatin: 210 mg, CIV 72 hours, administration method: continuous intravenous infusion, starting from the first day of each cycle; The subject underwent preoperative imaging evaluation and surgical indication evaluation one week after the end of the last medication before surgery. Subjects who still have indications for surgery after completing the two cycles before neoadjuvant therapy will receive surgical treatment within one week.

One week after surgery, the subjects began to receive a combination of trilaciclib chemotherapy (MAP regimen) and recombinant human endostatin adjuvant therapy for four cycles; Monitor adverse events (AE) throughout the entire study process and assess their severity level according to the guidelines listed in the National Cancer Institute (NCI) Common Terminology Standards for Adverse Events (CTCAE) version 5.0 or higher. Safety follow-up will be conducted on subjects receiving study treatment and early discontinuation of medication. The total survival of all subjects will be followed up until death, withdrawal of informed consent, or end of the study.

ELIGIBILITY:
Inclusion Criteria:

* 12 years old ≤ Age ≤ 50 years old, regardless of gender;
* Patients diagnosed by pathology and evaluated by surgeons as having unmetastased resectable osteosarcoma
* The patient's laboratory test meets the standards
* Cardiac echocardiography must meet the following criteria: Left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%).
* ECOG PS score 0-1 points;
* Women: All women with potential fertility must have a negative serum pregnancy test result during the screening period, and reliable contraceptive measures must be taken 3 months after signing the informed consent form and the last dose;
* Understand and sign the informed consent form.

Exclusion Criteria:

* Diagnosed as other malignant diseases outside of osteosarcoma within 5 years prior to initial administration (excluding curative basal cell carcinoma, squamous cell carcinoma of the skin, and/or radical resection of carcinoma in situ);
* Uncontrolled ischemic heart disease or clinically significant congestive heart failure (NYHA grade III or IV);
* Stroke or cardiovascular events within 6 months prior to enrollment;
* When screening, QTcF interval>480msec, for patients with implanted ventricular pacemakers, QTcF>500msec
* Previously received hematopoietic stem cell or bone marrow transplantation;
* Allergy to the investigational drug or its components;
* The researchers believe that it is not suitable to participate in this study.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade ≥ 3 neutropenia during chemotherapy treatment | 1-2 weeks after chemotherapy
  Is the number of neutrophils in the blood routine test lower than the ninth power of 1.0 * 10/L

SECONDARY OUTCOMES:
The incidence of grade 4 neutropenia during chemotherapy treatment | 1-2 weeks after chemotherapy
  Is the number of neutrophils in the blood routine test lower than the ninth power of 0.5 * 10/L
The occurrence of grade 3 or grade 4 thrombocytopenia during chemotherapy treatment | 1-3 weeks after chemotherapy
  Is the number of platelet in the blood routine test lower than the ninth power of 50 or 25 * 10/L
The incidence of grade 3 or 4 anemia during chemotherapy treatment | 1-3 weeks after chemotherapy
  Is the number of hemoglobin in the blood routine test lower than 80g/L

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
Shared mid-term data analysis report and final data analysis after patient enrollment
Supporting Information: CSR
Time Frame: August 2024 to June 2025